CLINICAL TRIAL: NCT02291419
Title: An Open Label, Randomized Study to Determine the Rate of Cardiovascular Events at 1 yr for Patients With Elevated Troponins Post Major Non-cardiac Surgery and the Impact of Ticagrelor vs Aspirin on the Occurrence of Cardiovascular Events
Brief Title: Study of Ticagrelor Versus Aspirin Treatment in Patients With Myocardial Injury Post Major Non-cardiac Surgery
Acronym: INTREPID
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment expectations were not met
Sponsor: The Cleveland Clinic (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Venu Menon, MD, FACC, FAHA, Director CICU, CEC-C5, Fellowship Program Cardiovascular Imaging, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCAZ-2014
Record Dates: First submitted 2014-11-05; First posted 2014-11-14 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Myocardial Injury
Keywords: ticagrelor; non-cardiac surgery; elevated troponin; myocardial injury
MeSH Terms: interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ticagrelor (Experimental): ticagrelor 90mg bid
  Interventions: Drug: ticagrelor
- aspirin (Active Comparator): Patients in the aspirin arm will receive aspirin 81 mg daily orally
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: ticagrelor — ticagrelor 90 mg bid
  Other Names: Brilinta
  Arms: ticagrelor
Drug: aspirin — aspirin 81 mg daily
  Other Names: Bayer, ASA
  Arms: aspirin

SUMMARY:
The purpose of this pilot study is to establish the rate of cardiovascular events in patients with elevated troponins levels after major, non-cardiac surgery and to evaluate the efficacy and safety of FDA approved study drug (ticagrelor) compared to aspirin in these patients.

Data from current studies suggest that myocardial injury detected by minor elevations in troponin levels within 3 days after non-cardiac surgery may occur in 10-24% of patients and is associated with an increased risk of mortality at 30 days and 1 year. There are no current guidelines for care of patients with elevated troponin levels in the absence of acute coronary syndrome. This study will assess if the increased risk of these patients is modifiable by an anti-platelet medication and evaluate the safety of this medication.

Patients will be randomized in an open label fashion to receive ticagrelor (anti-platelet medication) or 81 mg. aspirin. Patients will be followed on study treatment for 12 months, with the last contact at one month post treatment discontinuation.

DETAILED DESCRIPTION:
The objective of this pilot study is to establish the rate of cardiovascular events in patients with elevated troponins levels post major, non-cardiac surgery and to evaluate the efficacy and safety of ticagrelor treatment compared to aspirin in these patients.

Data from current studies suggest that myocardial injury detected by minor elevations in troponin levels within 3 days after non-cardiac surgery may occur in 10-24% of patients and is associated with an increased risk of mortality at 30 days and 1 year. There are no current guidelines for care of patients with elevated troponin levels in the absence of acute coronary syndrome (ACS) and it is not certain if this is a modifiable disease process. Ticagrelor is a direct, reversible inhibitor of the platelet P2Y12ADP-receptor. It has been shown to be superior to clopidogrel in the setting of ACS. The clinical benefit of treating patients with port-operative troponin elevation with antiplatelet agents remains unexplored. The short half-life of ticagrelor makes it favorable to use in this setting.

This is an open label, randomized, parallel group study comparing ticagrelor to aspirin in patients who experience troponin elevations post major non-cardiac surgery. Patients will be randomized in an open-label fashion to receive either ticagrelor 90 mg twice daily or aspirin 81 mg once daily. Patients will be followed for 13 months post randomization (12 months of treatment and a phone call 30 days after study drug discontinuation). The maximum duration of treatment will be 12 months.

Follow-up visits will occur at Month 1, Month 6, and Month 12. Phone calls will be made at Month 3, Month 9, and at 30 days after study drug discontinuation.

Up to 1000 patients with post-operative troponin elevation ≥2x ULN within first 7 postoperative days, will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before any study related procedures are performed.
2. A qualifying post-operative T or I troponin elevation (≥2x ULN of assay within 7 days of index surgery and during the index hospitalization).
3. Men and women ≥40 years of age if troponin elevation was identified as part of routine post-operative clinical care OR
4. Men and women ≥55 years of age if troponin elevation was identified post-operatively as part of screening for the study.
5. Undergone non-cardiac surgery requiring an overnight hospital stay.
6. Women of childbearing potential who are sexually active must have a negative pregnancy test at enrollment and agree to use adequate contraception from screening until 30 days after receiving the last dose of study drug.
7. Able to be randomized within 35 days following the index surgery.

Exclusion Criteria:

1. Post-operative ST-elevation Myocardial Infarction (STEMI).
2. Post-operative high-risk non-STEMI, defined as patients with elevated troponin with either:

   1. active Ischemic EKG changes (≥2 mm of ST-segment depression in at least 2 adjacent leads)
   2. ongoing hemodynamic instability thought to be ischemia mediated or
   3. persistent anginal symptoms.
3. Planned or urgent coronary angiography/revascularization.
4. A current or ongoing indication for dual antiplatelet therapy (DAPT) as determined by the patient's physician.
5. History of intracranial hemorrhage
6. Bleeding disorder or active bleeding that prevents ticagrelor or aspirin administration.
7. Taking any of the following medications at the time of randomization: vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxaban , fondaparinux, cilostazol, vorapaxar or LMWHs.
8. Renal dialysis.
9. Hepatic impairment with transaminase ≥3x ULN at time of randomization.
10. Known contra-indication for use of ticagrelor.
11. Estimated life expectancy of <1 year.
12. Enrolled in another ongoing drug or device research protocol
13. A definite non-ischemic explanation for troponin elevation, such as myocarditis or pulmonary embolism.
14. A documented hypersensitivity to aspirin.
15. Hypersensitivity to ticagrelor or any component of the product.
16. Neurological or ophthalmic surgery during the index hospitalization.
17. Patients taking strong CYP3A inhibitors and/or CYP3A inducers that cannot be stopped for the course of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venu Menon, MD, Principal Investigator — The Cleveland Clinic
Locations (24):
- United States (24):
  - University of South Alabama Health System, Mobile, Alabama
  - Arkansas Site Management Service, LLC, Little Rock, Arkansas
  - University of Florida College of Medicine - Jacksonville, Jacksonville, Florida
  - Florida Hospital Orthopaedic Institute and Fracture Care Center, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Central Georgia Heart Center, Macon, Georgia
  - Saint Vincent Medical Group, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - McLaren Bay Region, Bay City, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - New York University School of Medicine, New York, New York
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - VA Medical Center - Cleveland Louis Stokes, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - VA North Texas Health Care System, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Overlake Hospital Medical Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Background] POISE Study Group; Devereaux PJ, Yang H, Yusuf S, Guyatt G, Leslie K, Villar JC, Xavier D, Chrolavicius S, Greenspan L, Pogue J, Pais P, Liu L, Xu S, Malaga G, Avezum A, Chan M, Montori VM, Jacka M, Choi P. Effects of extended-release metoprolol succinate in patients undergoing non-cardiac surgery (POISE trial): a randomised controlled trial. Lancet. 2008 May 31;371(9627):1839-47. doi: 10.1016/S0140-6736(08)60601-7. Epub 2008 May 12. PMID 18479744
- [Derived] Horr S, Reed G, Menon V. Troponin elevation after noncardiac surgery: Significance and management. Cleve Clin J Med. 2015 Sep;82(9):595-602. doi: 10.3949/ccjm.82a.15076. PMID 26366956

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticagrelor | Aspirin
Started | 1 | 5
Completed | 0 | 0
Not Completed | 1 | 5
Not completed — Early study termination | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Aspirin | Total
Number analyzed (Participants) | 1 | 5 | 6
Age, Customized [Count of Participants; unit: Participants]
  > or = to 40 years | 1 | 5 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiovascular Events
Description: Time to first occurence of the composite of Cardiovascular Death, Non-fatal Myocardial Infarction, Coronary Revascularization or Non-fatal Stroke. The number of patients with events is reported.
Time Frame: up to 6 months. The planned duration of treatment was one year but the study was terminated after 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Aspirin
Number analyzed (Participants) | 1 | 5
Participants | 0 | 0

2. Secondary Outcome: Cardiovascular Death
Description: Time to first occurence of Cardiovascular death. The number of patients with events was reported.
Time Frame: Up to 6 months. The planned duration of treatment was one year but the study was terminated after 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Aspirin
Number analyzed (Participants) | 1 | 5
Participants | 0 | 0

3. Secondary Outcome: Non-fatal Myocardial Infarction or Coronary Revascularization
Description: Time to first occurence of Non-fatal myocardial infarction or coronary revascularization. The number of participants with events was reported.
Time Frame: up to 6 months. The planned duration of treatment was one year but the study was terminated after 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Aspirin
Number analyzed (Participants) | 1 | 5
Participants | 0 | 0

4. Secondary Outcome: All-cause Death
Description: Time to first occurence of All-cause death. The number of participants with events was reported.
Time Frame: up to 6 months. The planned duration of treatment was one year but the study was terminated after 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Aspirin
Number analyzed (Participants) | 1 | 5
Participants | 0 | 0

5. Secondary Outcome: Non-fatal Stroke
Description: Time to first occurence of Non-fatal stroke. The number of participants with events was reported.
Time Frame: up to 6 months. The planned duration of treatment was one year but the study was terminated after 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Aspirin
Number analyzed (Participants) | 1 | 5
Participants | 0 | 0

6. Other Pre Specified Outcome: The Number of Participants With Bleeding According to Bleeding Academic Research Consortium (BARC) Definitions
Time Frame: up to 6 months. The planned duration of treatment was one year but the study was terminated after 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor | Aspirin
Number analyzed (Participants) | 1 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored up to 6 months.
Arm/Group | Ticagrelor | Aspirin
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No